CLINICAL TRIAL: NCT05711472
Title: The Effect of Birth Ball Exercise on Labor Pain, Delivery Duration, Birth Comfort, and Birth Satisfaction
Acronym: BB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Seyhan Çankaya, Principal Investigator Seyhan Çankaya, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/1924
Record Dates: First submitted 2023-01-09; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Childbirth Problems; Labor Pain; Birth Disorder
Keywords: Birth pain; labor duration; birth comfort; birth satisfaction; birth ball
MeSH Terms: conditions — Labor Pain; Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Intervention Group Three different ball sizes, 55, 65 and 75 cm in diameter, were provided to the pregnant women, and the appropriate ball size was determined according to the height of the participant. In order for the pregnant woman to continue the balance exercises, they were allowed to sit on the round birth ball with their knees and hips at an angle of approximately 90°, with an upright spine. A birth ball of 55 cm was used for women between 150 and 160 cm in height, 65 cm for women between 160 and 170 cm, and 75 cm for women between 170 and 185 cm in height. Exercises with the round birth ball were guided by the researcher and the pregnant women performed the exercises in line with the guide.
  These are the movements performed with the round birth ball in 3 different positions: sitting (pelvic rocking movement, forward-backward and right-to-left rocking, forward supported sitting, and springing motion), kneeling, and squatting (ball hugging and pelvic rocking motion).
  Interventions: Other: birth ball exercise
- No Intervention (No Intervention): Control Group
  The followings were administered to the pregnant women in the Control Group after they were admitted to the hospital for delivery:
  * Information was given about the research,
  * Written consent was obtained,
  * Routine practices and care were provided in the delivery room (taking anamnesis, taking vital signs, demonstrating correct breathing techniques, ensuring freedom of movement)
  * Cervical changes were recorded on the partograph by vaginal examination,
  * EFM (Electronic Fetal Monitoring) was applied based on doctor's orders,
  * Fetal Heart Sound (FHS) was listened to every half hour and recorded on the partograph.

INTERVENTIONS:
Other: birth ball exercise — birth ball exercise used in childbirth
  Arms: Experimental

SUMMARY:
It has been reported that the birth ball has benefits such as decreasing the perception of labor pain, reducing the anxiety level, shortening the duration of the first stage of labor, increasing the satisfaction of birth, and facilitating the descent of the fetal head, but the literature is quite limited. So, this randomized controlled experimental study aimed to examine the effect of birth ball exercise on labor pain, delivery duration, birth comfort, and birth satisfaction.

DETAILED DESCRIPTION:
This randomized controlled experimental study aimed to examine the effect of birth ball exercise on labor pain, delivery duration, birth comfort, and birth satisfaction. The sample of the study consisted of 120 primiparous pregnant women presented to the delivery room between November 2021 and April 2022. Pregnant women were randomly assigned to the Intervention Group (IG, n=60) or the Control Group (KG, n=60). After the cervical dilatation reached at 4 cm, the pregnant women in the IG performed birth ball exercises, adhering to the birth ball guide created by the researcher. No intervention was made in the control group other than standard midwifery care practices.

A Personal Information Form,a Visual Analog Scale (VAS), the Childbirth Comfort Questionnaire (CCQ), a Labor and Postpartum Follow-up Form, and the Mackey Childbirth Satisfaction Rating Scale (MCSRS) were used for data collection. Women in both groups underwent VAS when cervical dilatation was 4 cm and 9 cm, and the CCQ was applied when dilatation was 8 cm. The MCSRS was administered two hours after delivery.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years or older;
* being in 37-42 weeks of pregnancy;
* having a singleton pregnancy;
* having a cervical dilatation of 1-4 cm;
* being primiparous;
* not having any complications that prevent vaginal delivery;
* not having any extremity problems for using the birth ball and performing activities;
* being able to speak and understand Turkish.

Exclusion criteria:

* Having maternal and fetal complications (oligohydramnios and polyhydramnios, placenta previa, preeclampsia, premature rupture of membranes, presentation anomalies, intrauterine growth retardation, fetal anomaly, intrauterine death, fetal macrosomia, fetal distress, etc.),
* getting pregnant by assisted reproductive techniques,
* electing cesarean section.

Exclusion criteria in the research process:

* To receive induction (oxytocin, prostaglandins, and misoprostol);
* having a cesarean delivery due to any complications;
* the baby admitted to the neonatal intensive care unit for any reason;
* receiving analgesics.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Personal information form before intervention | First 24 hours
  Assessed using personal information. This instrument includes questions about women's sociodemographic, obstetric and childbirth readiness characteristics.
Evaluation of birth | First 24 hours
  Birth Follow-up Form was used to evaluate labor. This Birth Follow-up form is evaluating; partograph, effacement-dilatation at first admission to the hospital, presence of amniotic sac at first admission, presence of episiotomy, time from active phase of labor until dilation is complete, time until the baby's head comes out after full dilation.
Evaluation of labor pain | First 24 hours
  Pain of pregnant women during labor was evaluated with Visual Analogue Scale (VAS). VAS scale, which would be applied to evaluate episiotomy pain in the postpartum period, was used to convert some values that cannot be measured numerically, and two-end definitions of the parameter to be evaluated are written at both ends of a 100 mm line. The participant was asked to indicate where his or her condition is suitable on this line by drawing a line or by placing a dot or pointing. "No pain" is written on one end and "very severe pain" on the opposite end; the participant was asked to mark the pain condition on this line.was used to convert some values that could not be measured numerically, and two-end definitions of the parameter to be evaluated are written at both ends of a 100 mm line.
Evaluation of Childbirth Comfort Questionnaire | First 24 hours
  Childbirth Comfort Questionnaire (CCQ) scales were applied to measure their comfort at the time of birth. The scale determines the comfort levels of women during childbirth. The real name of the scale is "Childbirth Comfort Questionnaire". The original scale consists of 14 items and is in a five-point Likert type. Each item is scored between 1-5.
Birth results information | Postpartum 1sth hours (after birth first 1 hour)
  Birth results information form evaluates; APGAR score at the 1st, 5th, and 10th minutes of the newborn; baby's gender.
Evaluation of Childbirth Satisfaction | Postpartum 1sth hours (after birth first 1 hour)
  Mackey Childbirth Satisfaction Rating Scale (MCSRS) evaluation to determine birth satisfaction form has been applied. The scale assesses women's satisfaction with the birth process. The scale consists of six 34-item subscales (nine items about self-satisfaction, two items about spouse's satisfaction, three items about baby's satisfaction, nine items about midwife-nurse satisfaction, eight items about doctor's satisfaction, three items about labor pain and labor. satisfaction). The scale is 5-point Likert type and is scored between 1 and 5. The lowest score in the scale is 32 and the highest score is 169, and as the total score increases, birth satisfaction also increases.

CONTACTS AND LOCATIONS:
Overall Officials: seyhan çankaya, PhD, Principal Investigator — Selcuk University
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No